CLINICAL TRIAL: NCT05924113
Title: Efficacy of Latin Dance for Promoting Wellbeing in Post Lung Transplant Recipients as Measured by Several Functional Measures, in the Outpatient Setting
Brief Title: A Study of Latin Dance for Post- Lung Transplant
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Teresa Padro, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-001508
Record Dates: First submitted 2023-06-20; First posted 2023-06-29 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Lung Transplant; Well-Being, Psychological
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Post-Lung Transplant (Experimental): Subjects that received a single or double lung transplants at Mayo Clinic Florida from 1/1/2020 to the present will participate in open sessions of Latin Dance over a 12-week period.
  Interventions: Behavioral: Latin Dance

INTERVENTIONS:
Behavioral: Latin Dance — Latin dance sessions that include a warm-up routine with music, two choreographed dances, and a cooldown routine with music.

SUMMARY:
The purpose of this research study is to see if participating in Latin dance for 12 sessions can improve wellbeing in several areas including balance, fear of movement, anxiety, depression and spirometry.

ELIGIBILITY:
Inclusion Criteria:

- Ambulatory with or without assisting devices (not on supplemental oxygen is not exclusionary), who have completed outpatient cardiopulmonary rehab and good pain control.

Exclusion Criteria:

- Tracheostomy, Hemodialysis, gastro-jejunal tubes, nasogastric tubes, wound vacs, chest tube, high levels of oxygen supplementation (mask vs nasal canula), recent falls.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in anxiety | Baseline, 12 weeks
  Measured using the General Anxiety Disorder 7-item (GAD 7) scale to assess severity of generalized anxiety disorder. Scoring is calculated by assigning scores of 0, 1, 2, and 3 to the response categories, respectively, of "not at all," "several days," "more than half the days," and "nearly every day." Total score for the seven items ranges from 0 to 21 where 0 is no anxiety, 1-4 is minimal anxiety, 5-9 is mild anxiety, 10-14 is moderate anxiety, and 15-21 is severe anxiety.
Change in depression | Baseline, 12 weeks
  Measured using the Patient Health Questionnaire 9-item (PHQ-9) scale to assess severity of depression. Scoring is calculated by assigning scores of 0, 1, 2, and 3 to the response categories, respectively, of "not at all," "several days," "more than half the days," and "nearly every day." Total score for the seven items ranges from 0 to 27 where 0 is no depression, 1-4 is minimal depression, 5-9 is mild depression, 10-14 is moderate depression, and 15-19 is moderately severe depression and 20-27 severe depression.
Change in Tampa Kinesophobia Scale | Baseline, 12 weeks
  Measured using the Tampa Scale for Kinesophobia 17-item scale to assess fear of movement. Scoring is calculated by assigning scores of 1, 2, 3, and 4 to the response categories, respectively, of "strongly agree," "disagree," "agree," and "strongly agree." Total score for the seventeen items ranges from 17 to 68. A score of 17 is the lowest possible score, and indicates no kinesiophobia or negligible. A score of 68 is the highest possible score and indicates extreme fear of pain with movement.

SECONDARY OUTCOMES:
Change in gait | Baseline, 12 weeks
  Measured using the Dynamic Gait Index 8-item scale to assess the likelihood of falling. Scoring is calculated by assigning scores of 0, 1, 2, and 3 to the response categories, respectively, of "severe impairment," "moderate impairment," "mild impairment," and "normal". Total score for the eight items ranges from 0 to 24 where 0 is the lowest level of function and 24 is the highest level of function.
Change in Forced Expiratory Volume in one second (FEV1) | Baseline, 12 weeks
  Measured by spirometry to determine the volume of air (in liters) exhaled in the first second during forced exhalation

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Padro, DNP, APRN, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials